CLINICAL TRIAL: NCT01445938
Title: An Open-label, Randomized Multicenter Study to Investigate the Anti-parasitic Activity, Pharmacokinetic and Safety of IM SAR97276A With Oral ACTs as Positive Control in Children Presenting With Symptomatic Plasmodium Falciparum Uncomplicated Malaria
Brief Title: Anti-parasitic Activity and Safety Assessment of SAR97276A in Children With Uncomplicated Malaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data Monitoring Committee recommendation
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDY11737; 2010-021398-36 (EudraCT Number); U1111-1118-0694 (Other: UTN)
Record Dates: First submitted 2011-09-26; First posted 2011-10-04 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Lumefantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Step 1 (SAR97276A od) (Experimental): 1 group of paediatric patients will receive 0.5 mg/kg SAR97276A administration once daily (od) for 3 days
  Interventions: Drug: SAR97276A
- Step 1 (SAR97276A bid) (Experimental): 1 group of paediatric patients will receive 0.25 mg/kg SAR97276A administration twice daily (bid) for 3 days
  Interventions: Drug: SAR97276A
- Step 1 (ACTs) (Active Comparator): 1 group of paediatric patients will receive arthemeter + lumefantrine (ACTs) bid for 3 days
  Interventions: Drug: arthemeter + lumefantrine (ACTs)
- Step 2 (SAR97276A) (Experimental): 1 or 2 groups of paediatric patients will receive SAR97276A once daily (od) or twice a day (bid) administration for 3 days (the choice of the od or bid regimen will be based on the results obtained in step 1)
  Interventions: Drug: SAR97276A
- Step 2 (ACTs) (Active Comparator): 1 group of paediatric patients will receive arthemeter + lumefantrine (ACTs) bid for 3 days
  Interventions: Drug: arthemeter + lumefantrine (ACTs)
- Step 3 (SAR97276A) (Experimental): 1 group of paediatric patients (2 to 11 years old) will receive: SAR97276A od or bid administration for 3 days (depending on results of step 1)
  Interventions: Drug: SAR97276A

INTERVENTIONS:
Drug: SAR97276A — Pharmaceutical form:solution for injection
  Route of administration: intramuscular
  Arms: Step 1 (SAR97276A bid); Step 1 (SAR97276A od); Step 2 (SAR97276A); Step 3 (SAR97276A)
Drug: arthemeter + lumefantrine (ACTs) — Pharmaceutical form:tablet
  Route of administration: oral
  Arms: Step 1 (ACTs); Step 2 (ACTs)

SUMMARY:
Primary Objective:

To assess the antiparasitic activity of intramuscular (IM) SAR97276A based on parasite reduction ratio at 72 hours in pediatric patients with uncomplicated malaria

Secondary Objectives:

* To assess the evolution of clinical signs and symptoms (including the need for a rescue therapy) in pediatric patients with uncomplicated malaria receiving SAR97276A with reference to Artemisinin-Based Combination Therapy (ACTs)
* To assess the pharmacokinetics profile of SAR97276A in pediatric patients with uncomplicated malaria
* To assess the safety profile of SAR97276A in pediatric patients with uncomplicated malaria
* To assess the pharmacokinetic-pharmacodynamic relationship of SAR97276A

DETAILED DESCRIPTION:
The total duration per patients will last approximately 28 ± 2 days broken down as follows:

* A screening phase up to 12-hours
* A 28 ± 2 days study period

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with symptomatic infection by Plasmodium falciparum microscopically confirmed in blood smear at Day-1 visit
* Fever (tympanic or rectal temperature ≥ 38 C) or documented history of fever within the last 24h
* Asexual parasitemia of ≥ 2 000 parasites/μL in blood smear at D-1 visit
* Signed Informed Consent Form by the parents or legal guardian
* Age: 12 to 17 years old for step 1
* Age: 2 to 11 years old for step 2 and step 3

Exclusion criteria:

* Participation in another clinical trial within the last 3 months or participation within a different cohort in this PDY11737 clinical trial or participation to previous trial with SAR97276
* Documented history of adequate treatment with antimalarials expected to be effective within the preceding 72 hours
* Severe concomitant disease (including concomitant febrile illnesses or infection)
* Any sign suggestive of severe malaria
* Severe malnutrition
* Asexual parasitemia: Plasmodium falciparum > 100,000 parasites/μL in blood smear at D-1 visit
* Previous treatment within 3 weeks prior to inclusion, and concomitant treatment with potent CYP3A4 inhibitors or CYP3A4 inducers or CYP2D6 substrates or potent CYP2D6 inhibitors
* Known serious adverse event reaction or hypersensitivity to Artemisinin-Based Combination Therapy (ACTs) or any contraindications from the positive control therapy (Artemisinin Combined Treatments) or warning/precaution of use as defined in the respective National Product Labeling
* Pregnant or breast-feeding women
* Women of childbearing potential not protected by effective contraceptive method of birth control, or not willing to use an effective contraceptive(s) method(s) for the duration of the study (e.g.: double barrier method), and/or who are unwilling or unable to be tested for pregnancy,
* CPK above 3 ULN,
* Underlying hepatobiliary disease or ALT>3 ULN.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Parasite Reduction Ratio (PRR) | at 72 hours

SECONDARY OUTCOMES:
Evolution of mean Parasitaemia over time (nb/µL) | every 6 hours from baseline up to 72 hours (day 4)
Evolution of mean Gametocytes count over time (nb/µL) | from baseline to end of study (day 28 ± 2)
Fever Clearance (time to reach Temperature < 38°C) | every 6 hours from baseline up to 72 hours (day 4)
General conditions improvement: mean total symptom score over time | every 6 hours from baseline up to 72 hours (day 4)
SAR97276 pharmacokinetic profile in plasma and blood | from baseline up to 12 hours after the last study drug intake on (Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Investigational Site Number 204001, Cotonou, Benin
- Investigational Site Number 854001, Ouagadougou, Burkina Faso
- Investigational Site Number 266001, Libreville, Gabon
- Investigational Site Number 404001, Kisumu, Kenya

REFERENCES:
- [Derived] Held J, Supan C, Salazar CLO, Tinto H, Bonkian LN, Nahum A, Sie A, Abdulla S, Cantalloube C, Djeriou E, Bouyou-Akotet M, Ogutu B, Mordmuller B, Kreidenweiss A, Siribie M, Sirima SB, Kremsner PG. Safety and efficacy of the choline analogue SAR97276 for malaria treatment: results of two phase 2, open-label, multicenter trials in African patients. Malar J. 2017 May 4;16(1):188. doi: 10.1186/s12936-017-1832-x. PMID 28472957